CLINICAL TRIAL: NCT00245505
Title: The Effect on Mucosal Healing With Pentasa Sachet 4g in Mild to Moderate Active Small Bowel Crohn´s Disease, Evaluated by Video Capsule Endoscopy After 6 and 12 Weeks Treatment. A Pilot Study
Brief Title: The Effect on Mucosal Healing With Pentasa Sachet in Mild to Moderate Active "Drug: Crohn's Disease"
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to lack of eligible patients
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE999907 CS004
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mesalazine (Mesalamine) — Pentasa (mesalazine) sachets 2 g morning + 2 g evening during 12 weeks treatment

SUMMARY:
The purpose of this study is to visualize the healing effect on mucosal lesions with Pentasa Sachet 4g in patients with mild to moderate active small bowel CD by video capsule endoscopy.

DETAILED DESCRIPTION:
The purpose of this study is to visualize the healing effect on mucosal lesions with Pentasa Sachet 4g in patients with mild to moderate active small bowel CD by video capsule endoscopy

ELIGIBILITY:
4.2 Inclusion Criteria

1. Patients who have signed the informed consent form
2. Patients with performed complete VCE < 7 days prior to inclusion and diagnosed clinically active mild to moderate small bowel CD and no stricture on previous examinations, as previously proven by barium small bowel follow through, enteroclysis and / or patency test capsule.
3. Patients between 18 - 70 years of age.

4.3 Exclusion Criteria

1. Patients with evidence of other forms of inflammatory small bowel bowel disease, idiopathic proctitis or infectious disease.
2. Patients with known small bowel strictures from previous examinations with for instance barium small bowel follow through, enteroclysis and / or patency capsule test.
3. Patients with pacemaker due to lack of VCE interaction data.
4. Patients who cannot undergo study procedures due to swallowing disorders.
5. Planned or actual pregnancy or lactation.
6. Women of child-bearing potential who are not using an effective method of contraception, in the opinion of the investigator.

8. Patients receiving maintenance treatment (p.o.) with total daily doses above 2.0g of sulphasalazine, mesalazine or 4-ASA, for 30 days prior to entry into the study.

9. Chronic use of non-steroidal anti-inflammatory drugs (oral and/or rectal routes) in 30 days prior to inclusion in the study (chronic use is defined as drug intake for a minimum of 3 consecutive days).

10. Intake of corticosteroids (oral and/or rectal routes) within the 30 days prior to enrolment in the study.

11. Patients receiving any immunosuppressive (azathioprine, 6-MP, etc) agents during 30 days prior to study enrolment.

12. Patients receiving any Crohn specific biological agents (TNF-alfa) during the last year prior to study enrolment.

13. Patients with any other disease or condition which may interfere with study assessments as judged by the investigator.

14. Alcoholism or drug addiction. 15. Patients participating or having participated in another clinical study in the previous 30 days.

16. Patients with severe renal/hepatic impairment (see section 5.6) as judged by the investigator.

17. Patients who are allergic to salicylate or 5-ASA derivatives. 18. Patients who are unlikely to comply with the protocol. 19. Any patient who has previously taken part in this study. 20. Patients who are unable to write or read local language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Mucosal changes, (measured as number, type and localization of small bowel mucosal lesions detected by VCE) from baseline (i.e. < 7 days prior to inclusion), and after 6 and 12 weeks´ treatment with 4g Pentasa Sachet | 12 weeks

SECONDARY OUTCOMES:
CDAI changes and laboratory changes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Department of Medicine, Malmö University Hospital, Malmo, Malmö, Sweden